CLINICAL TRIAL: NCT05287737
Title: Clinical Outcome After Total Pancreatectomy With Islet Autotransplantation
Acronym: TOPPER
Status: Enrolling by invitation | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Eelco JP de Koning, Prof. Eelco de Koning, Leiden University Medical Center
Other Study IDs: NL74838.058.21
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Islets of Langerhans Transplantation; Pancreatitis, Chronic; Diabetes Mellitus
Keywords: total pancreatectomy; autologous islet transplantation; TPIAT; beta-cell function; c-peptide
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Referred for Total pancreatectomy with islet autotransplantation: Followed up for up for 15 years after TPIAT.

SUMMARY:
A total pancreatectomy with islet autotransplantation (TPIAT) can be performed for a number of benign indications, such as chronic pancreatitis. In the current standard of treatment, after non-invasive, endoscopic efforts and other surgical options to relieve the pain, a total pancreatectomy is a last resort option. The pancreas is surgically removed during this procedure. Afterwards, the patient will have diabetes mellitus that is usually difficult to control with dependency on exogenous insulin administration. In TPIAT, a total pancreatectomy is followed by islet isolation from the resected pancreas and autotransplantation of these islets into the liver by means of a transhepatic intraportal islet infusion. Depending on the number and quality of islets, TPIAT may lead to full islet function so that no anti-hyperglycemic therapy is necessary or to partial islet function necessitating anti-hyperglycemic therapy. This can be only oral agents with reasonable islet function or complex insulin regimes with poor islet function. However, even with partial Islet function, glycemic control is easier with a lower risk of hypoglycemic events and diabetes-related complications, and an overall improvement of quality of life.

In this cohort, the endocrine function and glycemic variability will be monitored over time (up to 15 years). Additionally, pain scores, pain perception and central sensitization, quality of life, exocrine pancreatic insufficiency and diabetes-related stress will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for TPIAT or TPIAT performed since 2014
* Active and/or passive understanding of the Dutch language
* Willingness to wear a FGM or CGM device at least in the 2 weeks prior to TPIAT, first 3 months after TPIAT and for 2 weeks before yearly clinical visits.

Exclusion Criteria:

* Known malignancies of the pancreas

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for TPIAT or who have underwent TPIAT since 2014.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2047-03 (Estimated); Study Completion 2047-03 (Estimated)

PRIMARY OUTCOMES:
Pancreatic islet function | Up to 15 years
  AUC(0-120min) C-peptide during mixed meal tolerance test (MMTT)

SECONDARY OUTCOMES:
Pancreatic islet function | Up to 15 years
  Maximum C-peptide concentration during MMTT
Pancreatic islet function | Up to 15 years
  Difference in basal and maximum C-peptide concentration during MMTT
Glycemic control | Up to 15 years
  Time below range, time in range, time above range as determined by flash glucose monitoring (FGM) or continuous glucose measurement (CGM)
Glycemic control | Up to 15 years
  Standard deviation determined by FGM or CGM
Glycemic control | Up to 15 years
  HbA1c as determined in the blood and estimated by FGM or CGM
Glycemic control | Up to 15 years
  Insulin requirements (IU/kg/day)
Quality of life | Up to 15 years
  assessed by MOS Short Form 36 (SF-36) questionnaire
Quality of life | Up to 15 years
  assessed by EQ-5D questionnaire
Diabetes-related stress | Up to 15 years
  assessed by Problem Areas in Diabetes (PAID) questionnaire
Exocrine pancreatic insufficiency | Up to 15 years
  assessed by Pancreas Exocrine Insufficiency Questionnaire (PEI-Q)
Pancreas-related pain | Up to 15 years
  assessed by COMPAT-SF questionnaire
Pancreas-related pain | Up to 15 years
  assessed by Izbicki questionnaire
Pain perception and central sensitization | Baseline, MOS 6
  assessed by Quantitative Sensory Testing
Opioid usage | Up to 15 years
  Morphine Milligram equivalents
Frequency of surgical complications | Up to 15 years
  Early (<3 months) or late (>3 months)
Frequency of complications attributed to islet transplantation | Up to 15 years
Histological examination pancreas | After biopsy during islet isolation
  Degree of fibrosis, acinar cell atrophy, inflammation and nesidioblastosis

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Eelco de Koning, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided